CLINICAL TRIAL: NCT04315441
Title: Surveillance of Cardiovascular Risk Factors in Cameroonian Garrison
Status: Completed | Type: Observational
Sponsor: Support and Education Technic Centre (Other)
Responsible Party: Principal Investigator, Bienvenu BONGUE, Principal Investigator, Support and Education Technic Centre
Other Study IDs: UJM_UDD_01
Record Dates: First submitted 2020-03-12; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Risk Factor
Keywords: prevention; non-communicable disease; cardiovascular diseases; cardiovascular risk; soldiers
MeSH Terms: conditions — Noncommunicable Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Soldiers: any soldier who attended the Military Medical Center of Sector N°5 for the annual re-engagement medical visit during the period from January 1, 2017 to November 13, 2018.
  Interventions: Diagnostic Test: STEPS and AUDIT questionnaires
- Civilians: The civilian populations were recruited from two free cardiovascular risk factors screening campaigns carried out from January 04, 2017 to January 10, 2017 and from November 12, 2018 to November 18, 2018
  Interventions: Diagnostic Test: STEPS and AUDIT questionnaires

INTERVENTIONS:
Diagnostic Test: STEPS and AUDIT questionnaires — assessment was done according to World Health Organization STEPS manual for surveillance of risk factors of Non-communicable chronic diseases; and the Alcohol Use Disorders Identification Test. Five cardiovascular risk factors were assessed, smoking, harmful alcohol consumption, obesity/overweight, hypertension and diabetes. Cardiovascular risk was considered high in subjects with three or more cardiovascular risk factors.

SUMMARY:
Purpose: The objective of our study was to assess the cardiovascular risk of a Cameroonian military population and compare it to the cardiovascular risk of the neighboring civilian population.

Patients and methods: We will conduct a cross-sectional study that involved subjects aged from 18 to 58 years, recruited from October 2017 to November 2018 at the Fifth Military Sector Health Center in Ngaoundéré. Data collection and assessment was done according to World Health Organization STEPS manual for surveillance of risk factors of Non-communicable chronic diseases; and the Alcohol Use Disorders Identification Test. Five cardiovascular risk factors were assessed, smoking, harmful alcohol consumption, obesity/overweight, hypertension and diabetes. Cardiovascular risk was considered high in subjects with three or more cardiovascular risk factors. Univariates analysis and multivariate logistic regression were carried out according to their indications.

ELIGIBILITY:
Inclusion Criteria:

* agree to participate,
* had to be aged between 18 and 58 years old,
* representing ages of enrollment and retirement for Cameroonian soldiers respectively.

Exclusion Criteria:

-

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects of our study were recruited according to two methods at the Military Medical Center of Sector N°5 in Ngaoundere.
  Participation in the study was proposed to any soldier who attended the Military Medical Center of Sector N°5 for the annual re-engagement medical visit during the period from January 1, 2017 to November 13, 2018.
  The civilian populations were recruited from two free cardiovascular risk factors screening campaigns carried out from January 04, 2017 to January 10, 2017 and from November 12, 2018 to November 18, 2018. These campaigns were open to soldiers wishing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk factor | At inclusion
  evaluated by summing the participant's cardiovascular risk factors. The cardiovascular risk factors used for the cardiovascular risk assessment were smoking, excessive alcohol consumption (defined by an AUDIT score ≥ 8), overweight or obesity, hypertension, and diabetes. The cardiovascular risk was considered high if the subject had a combination of at least 3 cardiovascular risk factors.

SECONDARY OUTCOMES:
Smoking | At inclusion
  answering "yes" to the question do you smoke?
Alcoholism | At inclusion
  answering "yes" to the question do you consume alcohol?
Body mass index | At inclusion
  3 modalities was defined according to BMI. Underweight (BMI < 18.5 Kg/m2), normal weight (18 ≤ BMI < 25 Kg/m²), overweight (25 ≤ BMI < 30 Kg/m²), obesity (BMI ≥ 30 Kg/m²).
Systolic Blood Pressure (mmHg) | At inclusion
  Systolic blood pressure ≥ 140 mmHg or taking a hypotensive treatment.
Glycaemia (mmol/L) | At inclusion
  Fasting blood glucose ≥ 7 mmol/l or taking a hypoglycemic treatment
Diastolic Blood Pressure (mmHg) | At inclusion
  diastolic ≥ 90 mmHg or taking a hypotensive treatment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bell Ngan W, Essama Eno Belinga L, Essam Nlo'o ASP, Roche F, Goethals L, Mandengue SH, Bongue B. Surveillance of Cardiovascular Risk Factors in the Fifth Military Sector Health Center, Ngaoundere, Cameroon: Observational Study. JMIR Form Res. 2020 Nov 26;4(11):e18567. doi: 10.2196/18567. PMID 33242013